CLINICAL TRIAL: NCT00504803
Title: Mesenchymal Stem Cell Infusion as Prevention for Graft Rejection and Graft-versus-host Disease After Allogeneic Hematopoietic Cell Transplantation With Nonmyeloablative Conditioning: a Pilot Study
Brief Title: Mesenchymal Stem Cell Infusion as Prevention for Graft Rejection and Graft-versus-host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TJB0601
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Hematological Malignancies
Keywords: HCT, nonmyeloablative, mesenchymal stem cells, GVHD
MeSH Terms: conditions — Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MSC co-infusion with either HLA-mismatched PBSC or cord blood
  Interventions: Procedure: Mesenchymal stem cell infusion

INTERVENTIONS:
Procedure: Mesenchymal stem cell infusion — Infusion of mesenchymal stem cells on the same day as hematopoietic stem cell infusion.
  Other Names: Mesenchymal stem cells

SUMMARY:
Mesenchymal Stem Cell Infusion as Prevention for Graft Rejection and Graft-Versus-Host Disease After Allogeneic Hematopoietic Cell Transplantation With Nonmyeloablative Conditioning from HLA-mismatched PBSC or cord blood: a Pilot Study

ELIGIBILITY:
V.1. Patients

V.1.1. Diseases

Hematological malignancies confirmed histologically and not rapidly progressing:

* AML in CR;
* ALL in CR;
* CML unresponsive/intolerant to Imatinib but not in blast crisis;
* Other myeloproliferative disorders not in blast crisis and not with extensive myelofibrosis;
* MDS with < 5% blasts;
* Multiple myeloma;
* CLL;
* Non-Hodgkin's lymphoma (aggressive NHL should have chemosensitive disease);
* Hodgkin's disease.

V.1.2. Clinical situations

* Theoretical indication for a standard allo-transplant, but not feasible because:

  * Age > 55 yrs;
  * Unacceptable end organ performance;
  * Patient's refusal.
* Indication for a standard auto-transplant: perform mini-allotransplantation 2-6 months after standard autotransplant.

V.1.3. Other inclusion criteria

* Male or female; fertile female patients must use a reliable contraception method;
* Age < 75 yrs.
* Informed consent given by patient or his/her guardian if of minor age.

V.1.4. Exclusion criteria

* Any condition not fulfilling inclusion criteria;
* HIV positive;
* Terminal organ failure, except for renal failure (dialysis acceptable);
* Uncontrolled infection, arrhythmia or hypertension;
* Previous radiation therapy precluding the use of 2 Gy TBI;
* HLA-identical donor.

V.2. PBSC donors

V.2.1. Inclusion criteria

* Related to the recipient (sibling, parent or child) or unrelated;
* Male or female;
* Weight > 15 Kg (because of leukapheresis);
* Fulfills generally accepted criteria for allogeneic PBSC donation;
* Informed consent given by donor or his/her guardian if of minor age, as per donor center standard procedures.

V.2.2. Exclusion criteria

* Any condition not fulfilling inclusion criteria;
* HIV positive;
* Unable to undergo leukapheresis because of poor vein access or other reasons.

V.2.3. HLA matching

Related or unrelated donors who have 1-2 HLA mismatches, as either :

* One antigenic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1
* One allelic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1
* Two allelic mismatches at HLA-A or -B or -C or -DRB1 or -DQB1
* One antigenic mismatch + 1 allelic mismatch at HLA-A or -B or -C or -DRB1 or -DQB1.
* One antigenic mismatch at -DQB1 and one other antigenic mismatch at HLA-A or -B or -C or -DRB1

V.3. Cord blood unit

Banked cord blood units will be used if they fulfill the following criteria:

* No more than 2/6 HLA mismatches (antigenic mismatch at HLA-A or HLA-B or allelic mismatch at HLA-DRB1)
* > 2.5 x 107 TNC/kg
* Standard validation by FACT/Netcord criteria.

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Day-100 incidence of non-relapse mortality | 100 days

SECONDARY OUTCOMES:
1. Hematopoietic engraftment and graft rejection. 2. Incidence of grade II-IV and III-IV acute GVHD. 3. Immunologic reconstitution | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Baron, MD, PhD, Principal Investigator — CHU-ULg; Yves Beguin, MD, PhD, Principal Investigator — CHU-ULg; Chantal Lechanteur, PhD, Study Chair — CHU-ULg; Etienne Baudoux, MD, Study Chair — CHU-ULg; Evelyne Willems, MD, Study Chair — CHU-ULg
Locations (1):
- CHU Sart Tilman, Liège, Liege, Belgium

REFERENCES:
- [Derived] Baron F, Lechanteur C, Willems E, Bruck F, Baudoux E, Seidel L, Vanbellinghen JF, Hafraoui K, Lejeune M, Gothot A, Fillet G, Beguin Y. Cotransplantation of mesenchymal stem cells might prevent death from graft-versus-host disease (GVHD) without abrogating graft-versus-tumor effects after HLA-mismatched allogeneic transplantation following nonmyeloablative conditioning. Biol Blood Marrow Transplant. 2010 Jun;16(6):838-47. doi: 10.1016/j.bbmt.2010.01.011. Epub 2010 Jan 28. PMID 20109568